CLINICAL TRIAL: NCT01376219
Title: EU-COAST STUDY: European Cost of Asthma Treatment Economic Impact of Asthma Control
Brief Title: European Cost of Asthma Treatment
Acronym: EU-COAST
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113553
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
Keywords: GINA; direct / indirect costs; exacerbations; European; asthma control; Asthma Control Test (TM - QualityMetric Incorporated)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients entered in the study
  Interventions: Other: asthma control test

INTERVENTIONS:
Other: asthma control test — results of asthma control testing collected

SUMMARY:
The economic cost of asthma is considerable both in terms of direct medical costs (such as the cost of pharmaceuticals and hospital admissions) and indirect medical costs (such as time lost from work and premature death).

The costs of asthma depend on the severity of disease and the extent to which exacerbations are avoided. Moreover, poor control of asthma symptoms is a major issue that can result in adverse clinical and economic outcomes.

According to GINA guidelines, the goal of asthma treatment is to achieve and maintain asthma control. Such an objective can be reached in a majority of patients with a pharmacologic intervention strategy developed in partnership between the patient/family and the doctor. Validated measures for assessing asthma control score goals as continuous variables and provide numerical values to distinguish different levels of control. Among them, the Asthma Control Test (TM - QualityMetric Incorporated) is widely recognized. Few data exist on the relationship between asthma control and health care consumption.

Some models for predicting asthma costs have been proposed. However, these models only attempt to assess costs associated with medications and/or asthma exacerbations. Furthermore, in such studies, asthma control was not defined accordingly to current international criteria.

Considering the increasing interest of health authorities in reducing asthma associated costs and improving quality of care, it appears necessary to study the relationship between the cost and the level of control.

DETAILED DESCRIPTION:
A European observational retrospective bottom-up cost of illness study will be designed based upon a sample of patients with asthma. Investigators will be general practitioners.

They will have to enrol a sample of patients with asthma.

The level of asthma control will be evaluated with 2 methods:

* Firstly by using the auto-test Asthma Control Test (TM - QualityMetric Incorporated) which allows to assess the level of control on a 4-week period by distinguishing controlled and uncontrolled patients ;
* Secondly by using the GINA's asthma control criteria to measure the level of control in the last 3 months. The GINA classification will allow ranging patients in 3 groups (controlled, partly controlled and uncontrolled patients) and comprises a measure of lung function using a peak expiratory flow measurement (PEF) or a spirometric examination.

The study design will necessitate only one visit per patient with a retrospective data collection over a three-month period. This period is the maximum possible retrospective duration to avoid memory biases.

A questionnaire will be filled-up by the general practitioner. Data collected during the visit will be demographic data, medical history of patients, physician and paramedic's visits, treatment, diagnosis and lab tests, hospitalizations, rehabilitation, and absence from work during the last three months. A PEF or a spirometric result will be also requested. Patients will have to complete the Asthma Control test (TM - QualityMetric Incorporated) questionnaire. To assess the quality of life, patients will also have to complete the EQ-5D questionnaire.

As the time horizon of the asthma control concept is one month or shorter, the cost analysis will be first done taking into account this duration (the cost will be compared with the Asthma Control Test (TM - QualityMetric Incorporated) score), and secondly, on the three months period (the cost will be compared to the GINA's criteria).

To take into account seasonality, the overall population of patients will be enrolled in four quarterly waves. The data collection will therefore require one full year.

All the data collected will be centralized, captured and analyzed. Costing will be done using both societal and payer perspectives without any discounting. Results will be provided by period and by asthma control level and according to the patient profile (age, sex, etc.).

The number of patients needed to be enrolled was calculated taking into account the precision of the average cost estimate in the lower size group (i.e patients with optimal control) for each period in each country. In each country, at least 380 patients will be enrolled per wave to obtain a total population of 152 patients with optimal control. Overall, 3,040 will be enrolled all over the study year.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients, male or female aged ≥ 18 ;
* Patient diagnosed with asthma for at least 12 months and at least one antiasthmatic treatment in the last 12 months;
* Patient has read the information letter and the informed consent (if applicable).

Exclusion Criteria:

* Patient already included in this study;
* Patient who participated into a clinical trial during the last 6 months;
* Patient aged >=45 with an history of smoking of at least 20 packs-year;
* Patient with a chronic obstructive bronchopneumopathy
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with asthma for at least 12 months and at least one antiasthmatic treatment during the last 12 months
Sampling Method: Probability Sample
Enrollment: 2752 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
health care costs related to asthma according to the patients' asthma control level | 1 year

SECONDARY OUTCOMES:
Direct costs and indirect costs of consumed resources | 1 year
Costs directly associated with asthma care and costs associated with asthma complications (exacerbations); | 1 year
Healthcare costs related to asthma (by control) and concomitant diseases | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Barcelona, Spain